CLINICAL TRIAL: NCT05360576
Title: An Open-label, Randomized, 2-Period, Crossover Study to Assess the Comparative Pharmacokinetics of LSP-5415 and NuvaRing® in Healthy Adult Females
Brief Title: An Open-label, Randomized, 2-Period, Crossover, Pharmacokinetics Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lupin Research Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CVR-WH-201
Record Dates: First submitted 2022-01-21; First posted 2022-05-04 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy Prevention
MeSH Terms: interventions — etonogestrel; NuvaRing

STUDY DESIGN:
Intervention Model Description: All subjects will receive LSP-5415 (28 days) and NuvaRing (28 days) under fasted conditions. There will be a 28-day washout period after ring removal in Treatment Period 1 and ring insertion in Treatment Period 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LSP-5415 (etonogestrel/ethinyl estradiol vaginal ring) (Experimental): Test Product
  Interventions: Drug: LSP-5415 (etonogestrel/ethinyl estradiol vaginal ring); Drug: NuvaRing Vaginal Ring
- NuvaRing® (etonogestrel/ethinyl estradiol 11.7/2.7 mg) (Active Comparator): Reference Product
  Interventions: Drug: LSP-5415 (etonogestrel/ethinyl estradiol vaginal ring); Drug: NuvaRing Vaginal Ring

INTERVENTIONS:
Drug: LSP-5415 (etonogestrel/ethinyl estradiol vaginal ring) — To prevent pregnancy
  Other Names: LSP-5415
Drug: NuvaRing Vaginal Ring — To prevent pregnancy
  Other Names: NuvaRing

SUMMARY:
An Open-label, Randomized, 2-Period, Crossover Study to Assess the Comparative Pharmacokinetics of LSP-5415 and NuvaRing® in Healthy Adult Females

DETAILED DESCRIPTION:
This is an open-label, randomized-sequence, two-period, single-center, crossover, pharmacokinetic study in 40 healthy adult female subjects (18- 40 years). All subjects will receive LSP-5415 (28 days) and NuvaRing (28 days) under fasted conditions. There will be a 28-day washout period after ring removal in Treatment Period 1 and ring insertion in Treatment Period 2.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able, and willing, to sign Informed Consent Form prior to study participation in accordance with legal requirements.
2. Females (18 to 40 years of age, inclusive) without uncontrolled concomitant disease at Baseline Visit.
3. Have a regular menstrual cycle that is 24-32 days in duration.
4. Body Mass Index (BMI) of 18 kg/m2 to 30 kg/m2.
5. Will not be at risk for pregnancy, subjects must agree to consistently use reliable non-hormonal contraceptive methods (spermicide-coated condoms, male partner's sterilization via vasectomy, or sexual abstinence), or be in a same-sex relationship from screening through study completion, or be surgically sterilized by bilateral tubal ligation. -
6. Subjects must be in good physical and mental health as determined by vital signs, medical history.
7. Subjects must have a Blood Pressure reading in a sitting position, between 90-140 mmHg (systolic) and 50-90 mmHg (diastolic) and pulse rate between 50 and 100 bpm.
8. Be at least 3 months after a delivery or abortion.
9. Willing to abstain from vaginal products e.g., tampons, intravaginal medications etc. during the ring wear period for the study duration except water based vaginal lubricants/spermicides.

Exclusion Criteria:

1. Pregnancy, a positive serum ß-hCG pregnancy test at screening or lactation.
2. Use of tobacco- or nicotine-containing products (e.g., cigarette, pipe, cigar, chewing, vaping, nicotine patch, or nicotine gum) within 6 months prior to check-in on Day -1.
3. Have a history of cervical carcinoma or other carcinomas of the vagina or vulva.
4. Have a history of breast cancer or any hormonally sensitive cancer.
5. Subjects with abnormal pap smears that require colposcopic evaluations as defined by the fourth American Society of Colposcopy and Cervical Pathology (ASCCP) sponsored guidelines for management of cervical cancer abnormalities during the next 6 months are excluded until they have undergone colposcopic evaluation which has determined that a cervical procedure is not necessary during the 6 months following the colposcopy.
6. History of thrombophlebitis, venous or arterial thromboembolic diseases (thrombosis, pulmonary embolism, stroke or myocardial infarction).
7. Any known severe neurological, gastrointestinal, hepatic or other disease that might interfere with the intake of an investigational drug or any study condition.
8. Clinically relevant findings from serum biochemistry and hematology and HBsAg and C Virus/HlV serology as evaluated by the investigator.
9. Clinically relevant/significant electrocardiogram (ECG) findings.
10. Additional contraindications related to the use of ethinyl estradiol (EE), or hormonal contraceptives including women with a high risk of arterial or venous thrombotic diseases. Examples include women who are known to:

    1. Have cerebrovascular disease
    2. Have coronary artery disease
    3. Have thrombogenic valvular or thrombogenic rhythm diseases of the heart (for example, subacute bacterial endocarditis with valvular disease, or atrial fibrillation)
    4. Have inherited or acquired hypercoagulopathies
    5. Have uncontrolled hypertension
    6. Have diabetes mellitus with vascular disease
    7. Have headaches with focal neurological symptoms or migraine headaches with aura
11. History of migraine with focal neurological symptoms.
12. Known hereditary or acquired predisposition for venous and/or arterial thromboembolism (e.g., activated protein C [APC] resistance, anti-cardiolipin antibodies).
13. Less than 2 weeks remobilization after major surgery or prolonged immobilization
14. Alcohol, drug, or medicine abuse, or suspicion thereof.
15. Known allergy to any ingredient of the investigational drug.
16. Use of long-acting injectable or implant hormonal therapy. A washout period of 10 months and two regular cycles is required for long-acting injectable contraceptive therapy or implant hormonal therapy (e.g., depo-medroxyprogesterone) prior to the start of screening.
17. Use of hormonal or non-hormonal IUDs within 30 days prior to the start of screening.
18. Participation in another clinical trial at same time or within the preceding three months
19. Not fulfilling study specific requirements at screening.
20. Subjects desire to become pregnant during the Study.
21. Undiagnosed vaginal discharge/bleeding, vaginal lesions/ abnormalities or undiagnosed abnormal uterine bleeding. Subjects suspected of having a vaginal infection (e.g., chlamydia, gonococcus, yeast, trichomoniasis, or bacterial vaginosis, etc.) may be enrolled after treatment and subsequent negative test results; partner treatment is also recommended (as per treatment guidelines).
22. Regular intake or use of the following medication:

    1. any drugs that might interfere with the investigational drug.
    2. any hormonal preparation 30 days prior to the start of screening (except for treatment for thyroid disorders under control).
    3. any drugs known to induce liver enzymes (e.g., rifampicin, dexamethasone, barbiturates, anticonvulsants, St. John's Wort).
    4. any drugs known to inhibit CYP 3A4 (e.g. ketoconazole, verapamil, cimetidine, macrolides).
    5. any broad-spectrum antibiotics.
    6. use of Hepatitis C drug combinations containing ombitasvir/paritaprevir/ritonavir, with or without dasabuvir, due to potential for ALT evevations

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females of reproductive age
Enrollment: 40 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax) | 28 Days
  To assess the pharmacokinetics (PK) (Cmax) of etonogestrel (ENG) and ethinyl estradiol (EE) following LSP-5415 (28 days) and NuvaRing (28 days) administration.
Pharmacokinetics (Tmax) | 28 Days
  To assess the pharmacokinetics (PK) (Tmax) of etonogestrel (ENG) and ethinyl estradiol (EE) following LSP-5415 (28 days) and NuvaRing (28 days) administration.
Pharmacokinetics (AUC) | 28 Days
  To assess the pharmacokinetics (PK) (AUC) of etonogestrel (ENG) and ethinyl estradiol (EE) following LSP-5415 (28 days) and NuvaRing (28 days) administration.
Safety (Number of study subjects with treatment-emergent adverse events) | 3 months
  To assess the safety of LSP-5415 and NuvaRing in healthy adult female subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Mohope, Mumbai, India

IPD SHARING:
Plan to Share IPD: No